CLINICAL TRIAL: NCT00308802
Title: Noninvasive Monitoring to Predict Outcome in De Novo Kidney Transplant Recipients
Brief Title: Noninvasive Methods to Monitor Graft Survival in Kidney Transplant Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-01
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Transplant; Rejection; Kidney Disease; Kidney Failure; End Stage Renal Disease
MeSH Terms: conditions — Rejection, Psychology; Kidney Diseases; Renal Insufficiency; Kidney Failure, Chronic | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples may be retained
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Kidney transplantation — Participants in this study will have had a kidney transplant

SUMMARY:
The purpose of this study is to test noninvasive methods to monitor the health and condition of new kidneys in people who have received kidney transplants.

DETAILED DESCRIPTION:
Innovations in kidney transplantation have improved short-term outcomes for transplant patients. However, organ rejection remains as an important threat to the long-term survival of the transplanted organ. If clinicians could better monitor the condition of the organ after transplantation, they may be able to improve the chance of graft survival. Noninvasive ways to monitor the condition of the transplanted organ need to be developed and tested. This observational study will investigate whether certain blood and urine tests are useful in monitoring the health of transplanted kidneys.

This trial will involve 14 post-transplant study visits over the course of 2 years. A physical exam, medication history, adverse events assessment, and blood and urine collection will occur at all visits. Kidney biopsies will occur at study entry prior to transplantation and at Month 6, in adult participants only. Protocol biopsies are optional in the pediatric substudy group. Additional visits may be required if organ rejection is suspected.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for deceased donor or living donor kidney transplant
* Negative Crossmatch
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Clinically significant liver disease
* Other illnesses that, in the opinion of the investigator, may interfere with the study
* Recipient of multiple organ transplants
* Inability or unwillingness to comply with the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who are candidates for kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2006-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S. Heeger, MD, Study Director — Icahn School of Medicine at Mount Sinai; Donald Hricik, MD, Principal Investigator — University Hospitals Cleveland Medical Center; David Rush, MD, Principal Investigator — University of Manitoba at Winnipeg; Kenneth Newell, MD, Principal Investigator — Emory University; Richard Formica, MD, Principal Investigator — Yale University; Emilio Poggio, MD, Principal Investigator — The Cleveland Clinic; Barry Warshaw, MD, Principal Investigator — Emory-Children's Center; Enver Akalin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Patricia Birk, M.D., Principal Investigator — Children's Hospital of Winnipeg
Locations (9):
- United States (7):
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory Children's Center, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Mount Sinai School of Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
- Canada (2):
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Background] Kaplan B, Srinivas TR, Meier-Kriesche HU. Factors associated with long-term renal allograft survival. Ther Drug Monit. 2002 Feb;24(1):36-9. doi: 10.1097/00007691-200202000-00007. PMID 11805720
- [Background] Meier-Kriesche HU, Schold JD, Kaplan B. Long-term renal allograft survival: have we made significant progress or is it time to rethink our analytic and therapeutic strategies? Am J Transplant. 2004 Aug;4(8):1289-95. doi: 10.1111/j.1600-6143.2004.00515.x. PMID 15268730
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Result] Hricik DE, Nickerson P, Formica RN, Poggio ED, Rush D, Newell KA, Goebel J, Gibson IW, Fairchild RL, Riggs M, Spain K, Ikle D, Bridges ND, Heeger PS; CTOT-01 consortium. Multicenter validation of urinary CXCL9 as a risk-stratifying biomarker for kidney transplant injury. Am J Transplant. 2013 Oct;13(10):2634-44. doi: 10.1111/ajt.12426. Epub 2013 Aug 22. PMID 23968332
- See also: Click here for the Clinical Trials in Organ Transplantation (CTOT) public Web site — http://www.ctotstudies.org